CLINICAL TRIAL: NCT03974334
Title: Reducing Disparities in the Treatment of Hypertension Using the OWL mHealth Tool
Acronym: OWL-H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paula Gardiner (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institutes of Health (NIH) (NIH); University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor-Investigator, Paula Gardiner, Associate Professor, Associate Research Director, Medical Group Visit Program Director, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H00015619; 5U54HL143541-03 (NIH)
Record Dates: First submitted 2019-05-29; First posted 2019-06-04 (Actual); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Hypertension
Keywords: Blood Pressure, High
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: There are 2 cohorts taking part in the same intervention at 2 separate times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OWL-Hypertension 8 Wk Trial (Experimental): Two groups of thirteen participants will use the Our Whole Lives - Hypertension eHealth online tool for 8 weeks each, with baseline, midline, and follow-up data collected to determine any change due to the intervention.
  Interventions: Behavioral: OWL-Hypertension 8 Wk Trial

INTERVENTIONS:
Behavioral: OWL-Hypertension 8 Wk Trial — Our Whole Lives - Hypertension is an innovative online community and self-management program that provides access to stress reduction, mind-body techniques, nutrition, exercise, and peer support. OWL-H provides educational materials including videos of clinician-led talks (stress reactivity, nutrition, movement, etc.). OWL-H also provides subjects a facilitated community blog, private journal, peer support, and an extensive resource library. It will be tested by 26 patients with hypertension, to refine the platform based on patient feedback and outcomes.
  Other Names: Our Whole Lives - Hypertension

SUMMARY:
This is a one-year study. The study's primary outcome is successful improvement of the Our Whole Lives for Hypertension (OWL-H) online patient education platform, based upon participant use and focus group feedback, to deliver information on self-management of hypertension and other cardiac risk factors, and to encourage self-monitoring of blood pressure.

Specific Aim 1 - To pilot test the OWL-H platform for 8 weeks with 26 patients with hypertension (2 groups of 13) to refine its utility for home self-monitoring (number of times patients record home blood pressure and input this data onto OWL-H and engagement of self-management (i.e. # of logins, # of mind body sessions completed, # of times modules accessed each day)). Hypothesis 1: Eighty percent of patients will log in and record their blood pressures.

Specific Aim 2 - At the end of each group, hold a focus group to obtain information about: 1) the barriers and facilitators of using the OWL-H platform and using OWL-H to self-monitor blood pressure at home, 2) satisfaction with OWL-H, 3) how OWL-H helped with reduction of number of cardiac risk factors (e.g., smoking, eating habits, perceived stress, and amount of exercise and health-related quality of life).

DETAILED DESCRIPTION:
This is a one-year pre post clinical study. The study's primary outcome is successful improvement of the Our Whole Lives for Hypertension (OWL-H) online patient education platform, based upon participant use and focus group feedback, to deliver information on self-management of hypertension and other cardiac risk factors, and to encourage self-monitoring of blood pressure. We piloted online OWL-H platform for 8 weeks with 26 patients with hypertension to refine its utility for home self-monitoring. We also held a focus group to obtain information about: 1) the barriers and facilitators of using the OWL-H platform and using OWL-H to self-monitor blood pressure at home, 2) satisfaction with OWL-H, 3) how OWL-H helped with reduction of number of cardiac risk factors

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects of all races and ethnicities who are English-speaking adults over the age of 18 and who have a current diagnosis of hypertension.. OWL in currently only available in English.
* Subjects' physical and mental health status will be sufficient to be able to comprehend instructions and participate in the interventions.
* Subjects must be able to access computer technology (cellular phone, desktop, laptop) and the internet to utilize the online OWL-H.

Exclusion Criteria:

* Serious underlying systemic or co-morbid disease, including psychotic or manic symptoms, which preclude physical or cognitive ability to participate in the intervention.

The risk-benefit ratio of the interventions for these individuals may be potentially higher than acceptable.

* Active substance abuse, given that individuals who have active substance abuse pose a higher risk both to themselves and other members of the groups.
* Beginning new hypertension treatments in the past week or planning to begin new hypertension treatments in the next few weeks, or planning a major medical event in the next few weeks, which would interfere with accurately determining the effect of the intervention on impact in this study.
* Subjects who are pregnant will be not included in this study given that the risk-benefit ratio of this intervention may be higher than acceptable for these individuals due to the potential onset of non-study related gestational diabetes and/or gestational hypertension. Determination of pregnancy status will be based upon subject self-report.
* Subjects who are not willing to participate in the intervention or attend the group visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Gardiner, Associate Professor, Associate Research Director, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The data being collected is based on an intervention that is changing from cohort focus group to cohort focus group. It is also small sample size (n = 26) and only pilot data.

REFERENCES:
- [Background] Bartolome RE, Chen A, Handler J, Platt ST, Gould B. Population Care Management and Team-Based Approach to Reduce Racial Disparities among African Americans/Blacks with Hypertension. Perm J. 2016 Winter;20(1):53-9. doi: 10.7812/TPP/15-052. PMID 26824963
- [Background] Fang J, Yang Q, Ayala C, Loustalot F. Disparities in access to care among US adults with self-reported hypertension. Am J Hypertens. 2014 Nov;27(11):1377-86. doi: 10.1093/ajh/hpu061. Epub 2014 May 21. PMID 24847953
- [Background] Gardiner P, Dresner D, Barnett KG, Sadikova E, Saper R. Medical group visits: a feasibility study to manage patients with chronic pain in an underserved urban clinic. Glob Adv Health Med. 2014 Jul;3(4):20-6. doi: 10.7453/gahmj.2014.011. PMID 25105072
- [Background] Gardiner P, Lestoquoy AS, Gergen-Barnett K, Penti B, White LF, Saper R, Fredman L, Stillman S, Lily Negash N, Adelstein P, Brackup I, Farrell-Riley C, Kabbara K, Laird L, Mitchell S, Bickmore T, Shamekhi A, Liebschutz JM. Design of the integrative medical group visits randomized control trial for underserved patients with chronic pain and depression. Contemp Clin Trials. 2017 Mar;54:25-35. doi: 10.1016/j.cct.2016.12.013. Epub 2016 Dec 13. PMID 27979754
- [Derived] Gardiner P, McGonigal L, Villa A, Kovell LC, Rohela P, Cauley A, Rinker D, Olendzki B. Our Whole Lives for Hypertension and Cardiac Risk Factors-Combining a Teaching Kitchen Group Visit With a Web-Based Platform: Feasibility Trial. JMIR Form Res. 2022 May 16;6(5):e29227. doi: 10.2196/29227. PMID 35576575
- [Derived] Rohela P, Olendzki B, McGonigal LJ, Villa A, Gardiner P. A Teaching Kitchen Medical Groups Visit with an eHealth Platform for Hypertension and Cardiac Risk Factors: A Qualitative Feasibility Study. J Altern Complement Med. 2021 Nov;27(11):974-983. doi: 10.1089/acm.2021.0148. Epub 2021 Aug 5. PMID 34357790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from July-October of 2019 from Worcester, MA area adult primary care clinics, and either self-referred (via flyers and brochures placed around the clinics) or were referred by their primary care providers.They were then screened for eligibility, including a current diagnosis of hypertension in their EMR, and consented.
Groups:
- OWL-Hypertension 8 Wk Trial: Two groups of participants will use the Our Whole Lives - Hypertension mHealth online tool for 8 weeks each, with baseline, midpoint, and follow-up data collected to determine any change due to the intervention.
  OWL-Hypertension 8 Wk Trial: Our Whole Lives - Hypertension is an innovative online community and self-management program that provides access to stress reduction, mind-body techniques, nutrition, exercise, and peer support. OWL-H provides educational materials including videos of clinician-led talks (stress reactivity, nutrition, movement, etc.). OWL-H also provides subjects a facilitated community blog, private journal, peer support, and an extensive resource library. It will be tested by 26 patients with hypertension, to refine the platform based on patient feedback and outcomes.
Period: Overall Study
Arm/Group | OWL-Hypertension 8 Wk Trial
Started | 25
Completed | 24
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: One participant was lost to follow-up prior to Baseline data collection.
Arm/Group | OWL-Hypertension 8 Wk Trial
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 3
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 24
Blood Pressure Knowledge Questionnaire [Mean (Standard Deviation); unit: Scores on a scale] — The Blood Pressure Knowledge Questionnaire (BPKQ) was used to assess the participants' level of knowledge regarding common characteristics and risk factors of hypertension. It consists of 8 items covering topics like common symptoms, White Coat Syndrome, and the amount of salt consumed by the average American, with a mix of multiple choice (6 items) and true/false questions (2 items). The correct items are totaled, with a range of 1-8, and higher scores indicating more hypertension knowledge. The information needed to answer each item correctly was covered in OWL-H's curriculum.
  Scores on a scale | 5.58 (1.44)
Hypertension Self-Care Profile Self-Efficacy Instrument [Mean (Standard Deviation); unit: Scores on a scale] — The self-efficacy instrument of the Hypertension Self-care Profile (HTN-SCP-SE) used for this study consists of 20 items assessing the respondent's confidence on a scale of 1 (Not confident) to 4 (Very confident) to regularly engage in lifestyle habits that are recommended for patients with high blood pressure. It was developed and validated in 2014. The instrument results in a total confidence/self-efficacy score ranging from 20-80, with higher scores indicating higher levels of confidence in engaging in heart-healthy lifestyle habits.
  Scores on a scale | 63.67 (9.06)
Mediterranean Diet Questionnaire [Mean (Standard Deviation); unit: Scores on a scale] — The Mediterranean Diet Questionnaire (MDQ) consists of 14 yes-no items that assess participant's consumption of heart protective or harming foods. It was originally developed in Spain in 2004 to briefly assess adherence to a Mediterranean Diet and has been validated in multiple studies. Items assess the type of food eaten and whether the appropriate serving size is consumed, on a weekly basis. "Yes" responses are totaled, resulting in a score ranging from 0-14, with higher scores indicating a higher adherence to the Mediterranean Diet. Population: One participant did not fully complete this questionnaire at baseline, resulting in 23 rather than 24 participants assessed.
  Scores on a scale
    number analyzed (Participants) | 23
    (all) | 7.65 (2.19)
Blood Pressure Self-Monitoring (Self-Reported) [Mean (Standard Deviation); unit: Measurements/week] — To assess blood pressure self-monitoring pre-post, we first asked "Are you regularly (at least once per week) able to measure your blood pressure outside of your doctor appointments?". Those who said "yes" were then asked "How often, in a regular week, do you measure your blood pressure outside of your doctor appointments?" In their post-surveys, they were again asked to estimate their average weekly number of entries. Along with these self-report numbers, the OWL-H platform also keeps a log of every blood pressure entered by each participant across the 8 weeks. Population: Only 10 participants reported the ability to perform home self-monitoring of their blood pressure at Baseline.
  Measurements/week
    number analyzed (Participants) | 10
    (all) | 2.8 (1.31)

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Knowledge Questionnaire
Description: The Blood Pressure Knowledge Questionnaire (BPKQ) was used to assess the participants' level of knowledge regarding common characteristics and risk factors of hypertension. It consists of 8 items covering topics like common symptoms, White Coat Syndrome, and the amount of salt consumed by the average American, with a mix of multiple choice (6 items) and true/false questions (2 items). The correct items are totaled, with a range of 1-8, and higher scores indicating more hypertension knowledge. The information needed to answer each item correctly was covered in OWL-H's curriculum.
Time Frame: 8 Week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OWL-Hypertension 8 Wk Trial
Number analyzed (Participants) | 24
score on a scale | 6.13 (1.23)

2. Primary Outcome: Hypertension Self-Care Profile Self-Efficacy Instrument
Description: The self-efficacy instrument of the Hypertension Self-care Profile (HTN-SCP-SE) used for this study consists of 20 items assessing the respondent's confidence on a scale of 1 (Not confident) to 4 (Very confident) to regularly engage in lifestyle habits that are recommended for patients with high blood pressure. It was developed and validated in 2014. The instrument results in a total confidence/self-efficacy score ranging from 20-80, with higher scores indicating higher levels of confidence in engaging in heart-healthy lifestyle habits.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OWL-Hypertension 8 Wk Trial
Number analyzed (Participants) | 24
score on a scale | 65.54 (7.56)

3. Primary Outcome: Mediterranean Diet Questionnaire
Description: The Mediterranean Diet Questionnaire (MDQ) consists of 14 yes-no items that assess participant's consumption of heart protective or harming foods. It was originally developed in Spain in 2004 to briefly assess adherence to a Mediterranean Diet and has been validated in multiple studies. Items assess the type of food eaten and whether the appropriate serving size is consumed, on a weekly basis. "Yes" responses are totaled, resulting in a score ranging from 0-14, with higher scores indicating a higher adherence to the Mediterranean Diet.
Time Frame: 8 Weeks
Population: One participant did not fully complete this questionnaire at baseline, resulting in 23 rather than 24 participants assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OWL-Hypertension 8 Wk Trial
Number analyzed (Participants) | 23
score on a scale | 9 (1.68)

4. Secondary Outcome: Numbers of Time Blood Pressure Self-Monitoring Occurred During One Week
Description: To assess blood pressure self-monitoring pre-post, we first asked "Are you regularly (at least once per week) able to measure your blood pressure outside of your doctor appointments?". Those who said "yes" were then asked "How often, in a regular week, do you measure your blood pressure outside of your doctor appointments?" In their post-surveys, they were again asked to estimate their average weekly number of entries. Along with these self-report numbers, the OWL-H platform also keeps a log of every blood pressure entered by each participant across the 8 weeks.
Time Frame: 8 weeks
Population: One participant never entered a blood pressure reading in OWL-H.
Measure: Mean (Standard Deviation); unit: measurement per week
Arm/Group | OWL-Hypertension 8 Wk Trial
Number analyzed (Participants) | 23
measurement per week | 4.78 (1.90)

5. Secondary Outcome: Number of Time Blood Pressure Self-Monitoring on the OWL Platform Occurred Per Week
Description: Actual mean weekly entries of blood pressure readings in the OWL-H platform across the 8 weeks.
Time Frame: 8 Weeks
Population: One participant never entered a blood pressure reading in OWL-H.
Measure: Mean (Standard Deviation); unit: Measurements per week
Arm/Group | OWL-Hypertension 8 Wk Trial
Number analyzed (Participants) | 23
Measurements per week | 2.74 (2.02)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Any adverse event occurrences were captured through regular study staff and participants communications, as well as through provider/participant one-on-ones at the medical group visits held at Week 4 and 8 of the 8 week study.
Groups:
- OWL-Hypertension 8 Wk Trial: Two cohorts of participants will use the Our Whole Lives - Hypertension mHealth online tool for 8 weeks each, with baseline, midpoint, and follow-up data collected to determine any change due to the intervention.
  OWL-Hypertension 8 Wk Trial: Our Whole Lives - Hypertension is an innovative online community and self-management program that provides access to stress reduction, mind-body techniques, nutrition, exercise, and peer support. OWL-H provides educational materials including videos of clinician-led talks (stress reactivity, nutrition, movement, etc.). OWL-H also provides subjects a facilitated community blog, private journal, peer support, and an extensive resource library. It will be tested by 26 patients with hypertension, to refine the platform based on patient feedback and outcomes.
Arm/Group | OWL-Hypertension 8 Wk Trial
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
This feasibility study tested the OWL platform with hypertension patients in a regional medical center. Despite finding outcome improvements in lifestyle and self-management of HTN, a larger RCT is needed to assess for significant changes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT03974334/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT03974334/SAP_001.pdf
  • Informed Consent Form (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT03974334/ICF_002.pdf